CLINICAL TRIAL: NCT00448708
Title: Trial to Assess the Effectiveness of Maintaining Patency and Safety of the Vascular Wrap Paclitaxel-Eluting Mesh After Surgical Implantation With the Lifespan® ePTFE Vascular Graft in the Upper Extremity for Hemodialysis Vascular Access
Brief Title: Safety and Efficacy of Angiotech Vascular Wrap Paclitaxel-Eluting Mesh for Hemodialysis Vascular Access
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to an imbalance in graft infections between groups.
Sponsor: Angiotech Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012-VWAV06
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Results first posted 2011-11-17 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-10

CONDITIONS: Kidney Diseases; ESRD
Keywords: Hemodialysis Access
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vascular Wrap and Graft (Experimental): Lifespan® ePTFE Vascular Graft and Vascular WrapTM Paclitaxel-Eluting Mesh: The Lifespan® ePTFE Vascular Graft is implanted as an arteriovenous graft in an upper extremity to provide a hemodialysis access. The Vascular WrapTM Paclitaxel-Eluting Mesh is positioned on the vein and placed around the venous anastomosis to include both the toe and the heel of the anastomosis, and is sutured in place.
  Interventions: Device: Vascular Wrap Paclitaxel-Eluting Mesh; Device: Lifespan® ePTFE Vascular Graft
- Lifespan® ePTFE Vascular Graft (No Intervention): Lifespan® ePTFE Vascular Graft Only: The Lifespan® ePTFE Vascular Graft is implanted as an arteriovenous graft in an upper extremity to provide a hemodialysis access.
  Interventions: Device: Lifespan® ePTFE Vascular Graft

INTERVENTIONS:
Device: Vascular Wrap Paclitaxel-Eluting Mesh — 0.9 µg/mm^2 paclitaxel
  Other Names: Vascular Wrap; paclitaxel mesh
  Arms: Vascular Wrap and Graft
Device: Lifespan® ePTFE Vascular Graft — vascular graft
  Arms: Vascular Wrap and Graft
Device: Lifespan® ePTFE Vascular Graft — vascular graft
  Arms: Lifespan® ePTFE Vascular Graft

SUMMARY:
This is a multi-center clinical study in subjects requiring arteriovenous grafts in the upper extremity for hemodialysis access. All subjects will provide informed consent before undergoing any study procedures. The study will consist of multiple subject visits and telephone contacts during the 52 week study period. During the study period subjects must also maintain an appropriate hemodialysis schedule.

IDE Number: G060250

ELIGIBILITY:
Inclusion Criteria:

1. be ≥ 18 years of age;
2. if female of childbearing potential, provide evidence of a negative pregnancy test within 3 days prior to graft placement (Day -3 to Day 0);
3. be a candidate for a new end-to-side arteriovenous anastomosis graft placed in the upper extremity;
4. have an outflow vein of greater than or equal to 3 mm in diameter;
5. be able to effectively communicate with study personnel;
6. be considered by the physician to be available for subsequent visits;
7. be willing to comply with all aspects of the treatment and evaluation schedule over a 52 week duration;
8. allow representatives of the sponsor, designated CRO, Institutional Review Board (IRB), the Ethics Committee, and U.S. Food and Drug Administration (FDA) to review his/her relevant medical records;
9. sign and date an IRB-approved written informed consent prior to initiation of any study procedures, including screening procedures;
10. must agree to participate in protocol 014-VWAV07, a safety study to run consecutively for an additional 4 years or until Post-Market Approval (PMA), whichever is longer; and
11. have the Lifespan® ePTFE Vascular Graft successfully implanted.

Exclusion Criteria:

1. pregnant, breast-feeding, or female of childbearing potential who do not agree to remain abstinent or to use a contraceptive method during the study period. Non-childbearing potential is defined as either post-menopausal (amenorrheic for at least 1 year) or surgically sterile. Surgically sterile is defined as tubal ligation or the absence of the uterus and/or ovaries;
2. male of childbearing potential, who does not agree to remain abstinent or to use contraception to prevent fathering a child during the course of the study. Non-childbearing potential is defined as vasectomy or bilateral orchiectomy;
3. a central venous stenosis on the ipsilateral side is documented;
4. a hypercoagulable state is documented;
5. life expectancy is less than one year;
6. an organ transplant is expected within 6 months of test or control product (study products) placement;
7. hypersensitivity to any component of the study products or procedural materials or medications is known;
8. concurrently involved in another investigational study;
9. a study product being investigated by others has been received within 30 days prior to randomization in this trial;
10. the study product being studied in this trial has previously been received;
11. uncontrolled hypertension with systolic BP >200mmHg or diastolic BP >115mmHg is present at screening;
12. currently receiving chemotherapy or radiation therapy; or
13. placement of a new end-to-end arteriovenous anastomosis graft is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2007-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rui Avelar, MD, Study Chair — Angiotech Pharmaceuticals
Locations (33):
- United States (33):
  - Clinical Research Center, Birmingham, Alabama
  - Ladenheim, Inc., Fresno, California
  - Centinela Hospital, Inglewood, California
  - National Institute of Clinical Research, Los Angeles, California
  - USC CVTI - Healthcare Consultation II, Los Angeles, California
  - UCSD Medical Center, San Diego, California
  - Southern California Permanente Medical Group, San Diego, California
  - San Francisco VA Medical Center, San Francisco, California
  - Florida Research Network, LLC, Gainsville, Florida
  - Jacksonville Center for Clincal Research, Jacksonville, Florida
  - Discovery Medical Research Group, Ocala, Florida
  - Baptist Cancer Institute, Pensacola, Florida
  - Southeastern Urological Center, P.A, Tallahassee, Florida
  - University of South Florida- Research Foundation, Tampa, Florida
  - Cardiothoracic and Vascular Surgery Associates, Macon, Georgia
  - Renal Care Associates, Peoria, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - Washington County Hospital Association, Hagerstown, Maryland
  - Michigan Vascular Research Center, Flint, Michigan
  - Thoracic and Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Nephrology Associates P. C., Flushing, New York
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - Biomedical Research Alliance of New York, The Bronx, New York
  - BRANY - Montefiore Medical Center, The Bronx, New York
  - Rex Hospital, Raleigh, North Carolina
  - Clinical Research of Winston-Salem, Inc., Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Toledo, Toledo, Ohio
  - Health First Medical Group, Fort Worth, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Peripheral Vascular Associates, San Antonio, Texas
  - The Wisconsin Heart Hospital, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Vascular Wrap and Graft: Lifespan® ePTFE Vascular Graft and Vascular WrapTM Paclitaxel-Eluting Mesh
- Lifespan® ePTFE Vascular Graft: Lifespan® ePTFE Vascular Graft Only
Period: Overall Study
Arm/Group | Vascular Wrap and Graft | Lifespan® ePTFE Vascular Graft
Started | 112 | 110
Completed | 77 | 79
Not Completed | 35 | 31
Not completed — Death | 21 | 17
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Lost to Follow-up | 6 | 8
Not completed — not listed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vascular Wrap and Graft | Lifespan® ePTFE Vascular Graft | Total
Number analyzed (Participants) | 112 | 110 | 222
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 62 | 116
  >=65 years | 58 | 48 | 106
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (13.72) | 61 (15.58) | 63 (14.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 65 | 126
  Male | 51 | 45 | 96
Region of Enrollment [Number; unit: participants]
  United States | 112 | 110 | 222

OUTCOME MEASURES:

1. Primary Outcome: Time-to-loss of Target Site Primary Patency
Description: Subjects had primary patency at the target site from graft placement until an intervention on the target site occurred. The duration between graft implantation and graft abandonment due to loss of patency at the target site was the "time-to-loss of primary patency." Note: The study was halted early and therefore became underpowered to analyze efficacy as detailed in the protocol.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vascular Wrap and Graft | Lifespan® ePTFE Vascular Graft
Number analyzed (Participants) | 110 | 112
days | 130 [87 to 190] | 159 [86 to 227]

2. Secondary Outcome: Adverse Events
Description: adverse events with at least 5% incidence, reported as number of subjects experiencing the event (rather than total number of events). Adverse events were collected via subject querying at each visit and telephone contact, and by medical record review.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Vascular Wrap and Graft | Lifespan® ePTFE Vascular Graft
Number analyzed (Participants) | 110 | 112
participants
  Total Number of Adverse Events | 1451 | 1164
  Serious Adverse Events (deaths only) | 17 | 21

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Vascular Wrap and Graft | Lifespan® ePTFE Vascular Graft
Serious Adverse Events (participants affected / at risk) | 17/110 | 21/112
Other Adverse Events (participants affected / at risk) | 106/110 | 110/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vascular Wrap and Graft (N=110) | Lifespan® ePTFE Vascular Graft (N=112)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Cardiac arrest (Cardiac disorders) | 3 (3) | 2 (2) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Sepsis (Infections and infestations) | 1 (1) | 2 (2) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Septic shock (Infections and infestations) | 0 (0) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Dementia Alzhemier's type (Nervous system disorders) | 1 (1) | 0 (0) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Haemorrhage stroke (Nervous system disorders) | 0 (0) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Renal failure (Renal and urinary disorders) | 3 (3) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Hypotension (Vascular disorders) | 0 (0) | 2 (2) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
Death unknown cause (General disorders) | 2 (2) | 1 (1) — This adverse event resulted in death. Note: In this study, adverse events were never specifically captured as Serious Adverse Events. For this reason, no data other than "adverse events that resulted in death" are available for this category.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vascular Wrap and Graft (N=110) | Lifespan® ePTFE Vascular Graft (N=112)
Graft infection (Infections and infestations) | 32 (36) | 13 (14)
Anemia (Blood and lymphatic system disorders) | 15 (15) | 6 (6)
Leukocytosis (Blood and lymphatic system disorders) | 12 (12) | 5 (5)
Cardiac failure congestive (Cardiac disorders) | 6 (6) | 7 (7)
Tachycardia (Cardiac disorders) | 7 (7) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 8 (8)
Constipation (Gastrointestinal disorders) | 15 (15) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 14 (14) | 12 (12)
Nausea (Gastrointestinal disorders) | 30 (30) | 18 (18)
Vomiting (Gastrointestinal disorders) | 17 (17) | 9 (9)
Asthenia (General disorders) | 10 (10) | 8 (8)
Catheter related complication (General disorders) | 4 (4) | 6 (6)
Catheter site hemorrhage (General disorders) | 2 (2) | 7 (7)
Chest pain (General disorders) | 14 (14) | 10 (10)
Generalized oedema (General disorders) | 8 (8) | 2 (2)
Oedema peripheral (General disorders) | 26 (26) | 21 (21)
Pyrexia (General disorders) | 17 (17) | 12 (12)
Bacteraemia (Infections and infestations) | 8 (8) | 0 (0)
Catheter related infection (Infections and infestations) | 5 (5) | 6 (6)
Cellulitis (Infections and infestations) | 12 (12) | 7 (7)
Pneumonia (Infections and infestations) | 10 (10) | 13 (13)
Sepsis (Infections and infestations) | 13 (13) | 10 (10)
Urinary tract infection (Infections and infestations) | 12 (12) | 8 (8)
Excoriation (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Graft hemorrhage (Injury, poisoning and procedural complications) | 10 (10) | 4 (4)
Graft thrombosis (Injury, poisoning and procedural complications) | 41 (41) | 51 (51)
Wound dehiscence (Injury, poisoning and procedural complications) | 10 (10) | 0 (0)
Breath sounds abnormal (Investigations) | 12 (12) | 12 (12)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 4 (4) | 8 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 7 (7) | 14 (14)
Hypoglycemia (Metabolism and nutrition disorders) | 11 (11) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 (26) | 24 (24)
Dizziness (Nervous system disorders) | 10 (10) | 6 (6)
Headache (Nervous system disorders) | 12 (12) | 13 (13)
Hypoaesthesia (Nervous system disorders) | 7 (7) | 8 (8)
Unresponsive to stimuli (Nervous system disorders) | 7 (7) | 2 (2)
Anxiety (Psychiatric disorders) | 6 (6) | 2 (2)
Insomnia (Psychiatric disorders) | 9 (9) | 9 (9)
Mental status changes (Psychiatric disorders) | 7 (7) | 4 (4)
Anuria (Renal and urinary disorders) | 6 (6) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 10 (10)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Rales (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (9)
Erythema (Skin and subcutaneous tissue disorders) | 12 (12) | 3 (3)
Pruritis (Skin and subcutaneous tissue disorders) | 11 (11) | 8 (8)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6)
Hematoma (Vascular disorders) | 10 (10) | 8 (8)
Hypertension (Vascular disorders) | 13 (13) | 15 (15)
Hypotension (Vascular disorders) | 19 (19) | 23 (23)
Steal syndrome (Vascular disorders) | 8 (8) | 9 (9)
Thrombosis (Vascular disorders) | 11 (11) | 10 (10)
Venous stenosis (Vascular disorders) | 11 (11) | 10 (10)

LIMITATIONS AND CAVEATS:
Due to an observed imbalance in the number of graft infections, enrollment in the 1-year study 012-VWAV06 was suspended at the recommendation of the DSMC. Many of the planned efficacy analyses did not occur as a result of this suspension.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No